CLINICAL TRIAL: NCT07089485
Title: Impact of Anesthesia Alarm Volume on Mental Workload in Surgical Trainees: A Randomized Pilot Simulation Study
Brief Title: Impact of Anesthesia Alarm Volume on Mental Workload in Surgical Trainees
Acronym: ASLEC02
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-A01256-43
Record Dates: First submitted 2025-07-10; First posted 2025-07-28 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Surgical Procedures; Noise; Hearing Disorder; Mental Workload
Keywords: Noise/adverse effects; Cognition Disorders; Surgical procedures
MeSH Terms: conditions — Hearing Disorders; Cognition Disorders

STUDY DESIGN:
Intervention Model Description: This prospective interventional study will evaluate the impact of different noise levels in the operating room on surgeons' performance in simulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgical trainees group (Other): The study group consists of surgical trainees with limited experience in simulated surgery. They will perform multiple 15-minute surgical sequences in a controlled environment, where anesthesia alarm sound levels will vary between 64 and 75 dB(A). These sound levels will be randomized across the sequences to assess the impact of noise on their mental workload, concentration, and surgical performance.
  Interventions: Other: effects of sound

INTERVENTIONS:
Other: effects of sound — The surgical trainees will perform four 15-minute surgical sequences in a controlled environment, with varying sound levels (64, 67, 73, and 75 dB(A)) randomized across the sequences to assess the surgeons' responses.

SUMMARY:
Noise in hospital environments, particularly in operating rooms, poses challenges to both patient comfort and healthcare professionals' performance. Among the sources of noise, anesthesia monitoring alarms are essential for patient safety, yet no clear guidelines exist regarding their optimal sound level. Excessive alarm volume may increase distraction and cognitive load, especially for surgical trainees, potentially impairing their focus and performance during procedures. This randomized pilot interventional study aims to evaluate the impact of anesthesia alarm sound intensity on the mental workload of surgical trainees performing simulated surgeries. Participants will be randomly assigned to conditions with either an optimized alarm volume or a higher standard volume during simulated tasks. Cognitive load will be assessed using objective physiological measures such as heart rate variability and pupillometry, as well as subjective evaluations with tools like the NASA-TLX and SURG-TLX scales. The primary goal is to determine whether an optimized alarm sound level can reduce cognitive strain without compromising vigilance required for patient safety. Findings from this study are expected to provide evidence-based recommendations for auditory ergonomics in operating rooms, ultimately improving working conditions for surgical teams and enhancing both training and patient safety.

DETAILED DESCRIPTION:
Noise pollution in hospital environments, particularly within operating rooms (ORs), is a growing concern. It can impact not only the comfort and well-being of patients but also the cognitive performance and concentration of healthcare professionals. Among the various sources of noise, auditory alarms used in anesthesia monitoring are critical for patient safety. However, despite their importance, there are currently no established guidelines or regulations defining the optimal volume at which these alarms should be set.

Previous studies have examined the effects of background noise and music on surgical performance, with some showing that certain types of music can reduce stress or improve focus. However, the specific impact of anesthesia alarm sounds especially when they are excessively loud or frequent remains poorly understood. These alarms may distract surgical teams, particularly trainees, and contribute to increased cognitive load, potentially impairing performance during surgical procedures.

Cognitive load refers to the amount of mental effort being used in working memory. In the operating room, excessive cognitive load can hinder performance, decision-making, and reaction time, particularly in complex or high-pressure situations. Understanding how to manage and optimize environmental factors that influence mental workload is therefore essential, especially for surgical trainees still developing their skills.

This randomized pilot interventional study aims to investigate the effect of anesthesia alarm sound intensity on the mental workload of novice surgeons performing simulated procedures. By focusing on surgical trainees working on a high-fidelity simulator, we aim to create a controlled yet realistic environment to assess the cognitive impact of varying alarm volumes.

The study will compare two conditions: an optimized alarm sound level and a higher-level alarm sound (above ambient noise). Participants will be randomly assigned to one of these conditions during their simulated surgical tasks. The primary outcome is the cognitive load experienced by the trainees under each condition.

To comprehensively assess cognitive load, both objective and subjective tools will be used. Objective measures will include heart rate variability (HRV) and pupillometry two physiological indicators of stress and cognitive effort. Subjective cognitive load will be measured using validated scales such as the NASA Task Load Index (NASA-TLX) or its surgical adaptation, the SURG-TLX. These tools evaluate dimensions such as mental demand, effort, frustration, and performance.

By combining physiological data with subjective reports, the study seeks to capture a multidimensional understanding of how alarm noise affects surgical trainees. The ultimate goal is to determine whether reducing the intensity of auditory alarms while maintaining their effectiveness can minimize unnecessary cognitive strain and distraction during procedures.

The findings of this study are expected to inform future recommendations regarding auditory ergonomics in operating rooms. Establishing evidence-based guidelines for alarm sound levels could contribute to a safer, less stressful working environment for surgical teams. This is particularly important in the training context, where the balance between realism and cognitive manageability is crucial for learning and performance.

In conclusion, this pilot study addresses a critical and underexplored aspect of the surgical environment: the cognitive impact of anesthesia alarm noise. By evaluating its effects on novice surgeons, the research aims to promote better alarm management strategies, improve working conditions, and ultimately enhance both patient safety and surgical education.

ELIGIBILITY:
Inclusion Criteria:

* Surgical residents or experienced surgeons;
* Surgeons with normal hearing;
* Surgeons capable of performing surgical sutures (regardless of skill level);
* Surgeons able and willing to follow all study procedures according to the protocol;
* Surgeons who have understood, signed, and dated the informed consent form provided on the day of enrollment.

Exclusion Criteria:

* Surgeons undergoing beta-blocker treatment;
* Surgeons with known cardiac pathology;
* Surgeons who do not consent to participate in the study;
* Surgeons with known hearing problems;
* Surgeons who fail the hearing test;
* Surgeons who worked on-call or night shifts during the night before the evaluation day.
* Surgical trainees at the Lorraine Cancer Institute.
* Adults under legal protection (guardianship, curatorship, or legal supervision);Persons deprived of liberty;Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Impact of the optimal sound intensity level during a surgical procedure | From inclusion (baseline) to 6 months post-inclusion
  Assessment of heart and respiratory rate variability parameters

SECONDARY OUTCOMES:
Interference with the surgical procedure | From inclusion (baseline) until the end of the surgical procedure
  Measurement using the SURG-TLX (Surgical Task Load Index) questionnaire
Mental workload of the surgical trainee | From inclusion (baseline) until the end of the surgical procedure
  Measurement using the SURG-TLX scale.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric MARCHAL, Pr., Principal Investigator — Institut de Cancérologie de Lorraine; Nour Mammari Halabi, PhD., Study Chair — Institut de Cancérologie de Lorraine

IPD SHARING:
Plan to Share IPD: No
At this time, the individual participant data (IPD) will not be shared due to concerns regarding participant privacy and confidentiality, as well as institutional policies restricting data sharing.

REFERENCES:
- [Background] Roche TR, Said S, Braun J, Maas EJC, Machado C, Grande B, Kolbe M, Spahn DR, Nothiger CB, Tscholl DW. Avatar-based patient monitoring in critical anaesthesia events: a randomised high-fidelity simulation study. Br J Anaesth. 2021 May;126(5):1046-1054. doi: 10.1016/j.bja.2021.01.015. Epub 2021 Apr 8. PMID 33879327
- [Background] Torabizadeh C, Yousefinya A, Zand F, Rakhshan M, Fararooei M. A nurses' alarm fatigue questionnaire: development and psychometric properties. J Clin Monit Comput. 2017 Dec;31(6):1305-1312. doi: 10.1007/s10877-016-9958-x. Epub 2016 Nov 15. PMID 27848141
- [Background] Way TJ, Long A, Weihing J, Ritchie R, Jones R, Bush M, Shinn JB. Effect of noise on auditory processing in the operating room. J Am Coll Surg. 2013 May;216(5):933-8. doi: 10.1016/j.jamcollsurg.2012.12.048. Epub 2013 Mar 18. PMID 23518255
- [Background] Whitham MD, Casali JG, Smith GK, Allihien AL, Wright BW, Barter SM, Urban AR, Dudley DJ, Fuller RR. Noise in cesarean deliveries: a comprehensive analysis of noise environments in the Labor and Delivery operating room and evaluation of a visual alarm noise abatement program. Am J Obstet Gynecol MFM. 2023 May;5(5):100887. doi: 10.1016/j.ajogmf.2023.100887. Epub 2023 Feb 11. PMID 36781121
- [Background] Schmid F, Goepfert MS, Kuhnt D, Eichhorn V, Diedrichs S, Reichenspurner H, Goetz AE, Reuter DA. The wolf is crying in the operating room: patient monitor and anesthesia workstation alarming patterns during cardiac surgery. Anesth Analg. 2011 Jan;112(1):78-83. doi: 10.1213/ANE.0b013e3181fcc504. Epub 2010 Oct 21. PMID 20966440
- [Background] Katz JD. Noise in the operating room. Anesthesiology. 2014 Oct;121(4):894-8. doi: 10.1097/ALN.0000000000000319. No abstract available. PMID 24878496
- [Background] Lamotte AS, Essadek A, Shadili G, Perez JM, Raft J. The Impact of Classroom Chatter Noise on Comprehension: A Systematic Review. Percept Mot Skills. 2021 Jun;128(3):1275-1291. doi: 10.1177/00315125211005935. Epub 2021 Mar 27. PMID 33775178
- [Background] Fu VX, Oomens P, Sneiders D, van den Berg SAA, Feelders RA, Wijnhoven BPL, Jeekel J. The Effect of Perioperative Music on the Stress Response to Surgery: A Meta-analysis. J Surg Res. 2019 Dec;244:444-455. doi: 10.1016/j.jss.2019.06.052. Epub 2019 Jul 18. PMID 31326711
- [Background] El Boghdady M, Ewalds-Kvist BM. The influence of music on the surgical task performance: A systematic review. Int J Surg. 2020 Jan;73:101-112. doi: 10.1016/j.ijsu.2019.11.012. Epub 2019 Nov 22. PMID 31760139
- [Background] Oomens P, Fu VX, Kleinrensink GJ, Jeekel J. The effect of music on simulated surgical performance: a systematic review. Surg Endosc. 2019 Sep;33(9):2774-2784. doi: 10.1007/s00464-019-06868-x. Epub 2019 May 28. PMID 31140001